CLINICAL TRIAL: NCT06992726
Title: Mechanisms of n-3 Polyunsaturated Fatty Acids Promoting White Fat Beige Coloration to Improve Obesity With Cognitive Impairment by Regulating Intestinal Bacteriophages and Their Metabolites
Brief Title: Improvement of Fish Oil in Obesity With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weiwei Ma (Other)
Responsible Party: Sponsor-Investigator, Weiwei Ma, professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Z2023SY126
Record Dates: First submitted 2025-05-05; First posted 2025-05-28 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Mild Cognitive Impairment
MeSH Terms: conditions — Obesity; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator)
  Interventions: Other: Placebo intervention
- Fish oil intervention group (Experimental)
  Interventions: Dietary Supplement: Fish oil intervention

INTERVENTIONS:
Dietary Supplement: Fish oil intervention — The diet was based on the principles of a balanced diet, and subjects in this group were additionally supplemented with n-3 PUFA (provided as 1.36 g fish oil capsules), with the rest of the intervention being the same as in the control group.
  Arms: Fish oil intervention group
Other: Placebo intervention — Diet based on the principles of a balanced diet, taking placebo capsules with the same appearance and odor as the fish oil capsules.
  Arms: control group

SUMMARY:
Eighty-eight patients with obesity with mild cognitive impairment（MCI） from the Multicenter Nutrition and Chronic Disease Cohort, who met the inclusion and exclusion criteria, were selected as study subjects and randomly divided into 2 groups, i.e., the placebo group and the n-3 PUFA intervention group. Subjects in the intervention group were given supplemental n-3 PUFA (supplied in 1.36 g fish oil capsules); the placebo group took placebo (1.36 g/d), and the intervention period was 12 consecutive months. General information, dietary intake, body composition, exercise, overall cognitive function and multidimensional cognitive function, abundance of Mycobacterium avium and its metabolites acetic acid and propionic acid content, beige adiposity markers, inflammation-related factors, and lipid metabolism were collected at baseline, at the end of 6 months and at the end of 12 months of the intervention, respectively, and the adherence of the two groups of subjects was also assessed. To analyze the effects of n-3 PUFA intervention on cognitive function in patients with obesity with MCI and to explore the possible mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of obesity and MCI;
* Age between 35 and 80 years old;
* No dieting or stop dieting in the last 3 months, no fish oil supplements, or willing to stop self-administration of fish oil 3 months before the intervention;
* Voluntarily participate in the program with informed consent, and sign the informed consent form.

Exclusion Criteria:

* Those with neuropsychiatric disorders such as stroke, epilepsy, or schizophrenia;
* Those with cognitive impairment caused by depression, thyroid disease, traumatic brain injury, drug or alcohol intoxication;
* Those with a history of cerebrovascular disease or cognitive impairment caused by severe cardiac, hepatic, pulmonary, or renal impairment;
* Those who are complete vegetarians and are unable to comply with the balanced dietary pattern;
* Those who suffer from severe angina pectoris, asthmatic bronchitis, severe infections , systemic lupus erythematosus, malignant tumors, and other diseases that may affect one's dietary habits and life;
* Coeliac disease with lipid malabsorption.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Height, Waist | Baseline, 6 months, 12 months
  Measurement of the subject's height and waist circumference using a tape measure.
weight | Baseline, 6 months, 12 months
  The weight of the subjects was measured using a weighing scale.
Total Body Water | Baseline, 6 months, 12 months
  Measuring Total Body Water (L) with the InBody Body Composition Analyzer.
body protein, inorganic salts, and body fat | Baseline, 6 months, 12 months
  Measurement of body protein, inorganic salts, and body fat using the InBody Body Composition Analyzer (kg)
Appendicular skeletal muscle mass index | Baseline, 6 months, 12 months
  Skeletal muscle mass of the extremities is the sum of the muscle mass of both upper and lower extremity skeletal muscles, which was measured using a body composition meter. The appendicular skeletal muscle mass index (ASMI) is the mass of the skeletal muscles of the extremities divided by the square of the height (kg/m2).
Cognitive function assessment | Baseline, 6 months, 12 months
  Cognitive function was assessed using the Montreal Cognitive Assessment (MoCA) scale, which is a 30-point scale that includes multiple dimensions of cognitive functioning, including visuospatial and executive functioning, naming, memory, attention, language, abstraction, delayed recall, and orientation.
  The MCI diagnostic criteria were: <6 years of education, MoCA score ≤19; >7 years of education but ≤12 years, MoCA ≤22; >12 years of education, MoCA ≤24.
Dietary composition | Baseline
  The food frequency questionnaire (FFQ) was used for the survey assessment. With reference to the FFQ questionnaire used in the Nutrition and Health Status Survey of Chinese Residents, a total of 72 food inquiry entries in 11 food groups were included, with a focus on n-3 PUFA-rich foods, as well as the intake of edible oils and condiments. Auxiliary survey tools such as the Retrospective Dietary Survey Auxiliary Atlas were used to help respondents recall. The Standardized Version of the Chinese Food Composition Table (6th Edition) was used to calculate the energy and nutrient intake of the population, including the intake of dietary fatty acids.
Dietary Inflammation Index | Baseline
  The dietary inflammatory index (DI) for each dietary component/nutrient was calculated separately for each individual based on the mean and standard deviation of the per capita daily intake of each dietary component or nutrient and the corresponding dietary effect index of each component.If a food increases the level of pro-inflammatory factors or decreases the level of anti-inflammatory factors, it is labeled as "+1" for a pro-inflammatory effect; conversely, it is assigned "-1" for an anti-inflammatory effect. If there was no significant change in inflammatory markers, "0" was assigned as no pro/anti-inflammatory effect. The final DI score for each food was accumulated to obtain an overall dietary DI score for the individual; the higher the total DI score, the greater the pro-inflammatory effect of the diet, and conversely, the greater the anti-inflammatory effect.
Species and abundance of intestinal flora | Baseline, 6 months, 12 months
  Detection Methods:Fecal flora was detected by designing and amplifying sequences specific to B. anthropophilus and then applying RT-qPCR.
Metabolite levels of intestinal flora | Baseline, 6 months, 12 months
  HPLC-MS/MS
Plasma inflammatory factor levels | Baseline, 6 months, 12 months
  High-Throughput Liquid Protein Chip
Erythrocyte Membrane n-3 PUFA Levels | Baseline, 6 months, 12 months
  Gas Chromatography
Plasma Beige Lipid Marker Levels | Baseline, 6 months, 12 months
  Double antibody sandwich ELISA
Fecal Akkermansia abundance | Baseline, 6 months, 12 months
  qPCR
Fecal Amuc_1100 expression levels | Baseline, 6 months, 12 months
  Fecal Amuc_1100 mRNA expression was detected using Realtime-PCR.
Detection of signaling pathway related indicators of plasma fat metabolism | Baseline, 6 months, 12 months
  Enzyme colorimetric method
Levels of lipopolysaccharide | Baseline, 6 months, 12 months
  Enzyme colorimetric method
Plasma lipid oxide concentrations | Baseline, 6 months, 12 months
  LC-MS/MS
Levels of fatty acid synthetase | Baseline, 6 months, 12 months
  Enzyme colorimetric method

SECONDARY OUTCOMES:
Blood lipids | Baseline, 6 months, 12 months
  Enzyme colorimetric method
Fasting blood glucose | Baseline, 6 months, 12 months
  Hexokinase method

CONTACTS AND LOCATIONS:
Overall Officials: Ruiqi Mu, Principal Investigator — Capital Medical University

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT06992726/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT06992726/ICF_001.pdf